CLINICAL TRIAL: NCT01914432
Title: A Double-blind, Randomized, Multi-center Phase III Clinical Trial to Investigate the Safety and Efficacy Between YH16410 Versus Rosuvastatin and Telmisartan Monotherapies in Patients With Hypertension and Hyperlipidemia
Brief Title: Efficacy and Safety Study of YH16410 Versus Rosuvastatin and Telmisartan Monotherapies in Patients With Hypertension and Hyperlipidemia
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Yuhan Corporation (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: YH16410-301
Record Dates: First submitted 2013-07-30; First posted 2013-08-02 (Estimated); Last update posted 2014-07-08 (Estimated); Status verified 2014-07

CONDITIONS: Hyperlipidemia; Hypertension
MeSH Terms: conditions — Hyperlipidemias; Hypertension | interventions — Rosuvastatin Calcium; Telmisartan

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (4):
- YH16410 (Experimental): PO, Once Daily, 8 weeks
  Interventions: Drug: YH16410; Drug: Rosuvastatin placebo; Drug: Telmisartan placebo
- Rosuvastatin (Active Comparator): PO, Once Daily, 8 weeks
  Interventions: Drug: Rosuvastatin; Drug: YH16410 placebo; Drug: Telmisartan placebo
- Telmisartan (Active Comparator): PO, Once Daily, 8 weeks
  Interventions: Drug: Telmisartan; Drug: YH16410 placebo; Drug: Rosuvastatin placebo
- Placebo (Placebo Comparator): PO, Once Daily, 8 weeks
  Interventions: Drug: YH16410 placebo; Drug: Rosuvastatin placebo; Drug: Telmisartan placebo

INTERVENTIONS:
Drug: YH16410
  Arms: YH16410
Drug: Rosuvastatin
  Arms: Rosuvastatin
Drug: Telmisartan
  Arms: Telmisartan
Drug: YH16410 placebo
  Arms: Placebo; Rosuvastatin; Telmisartan
Drug: Rosuvastatin placebo
  Arms: Placebo; Telmisartan; YH16410
Drug: Telmisartan placebo
  Arms: Placebo; Rosuvastatin; YH16410

SUMMARY:
To evaluate efficacy and safety of YH16410 versus rosuvastatin and telmisartan monotherapies in patients with hypertension and hyperlipidemia

ELIGIBILITY:
Inclusion Criteria:

* Signed Informed Consent
* Men and women ≥ 19 years of age
* Subject who has one of 3 conditions classified by Cardiovascular Risk Factors, 10-Year Risk, Blood Pressure, LDL-C, TG, Coronary Artery Disease and Equivalent

Exclusion Criteria:

* Females who are pregnant, breastfeeding, or of childbearing potential, unwilling to practice adequate contraception throughout the study.
* Other exclusions applied

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 210 (Actual)
Dates: Start 2013-11; Primary Completion 2014-06 (Actual); Study Completion 2014-06 (Actual)

PRIMARY OUTCOMES:
Change in Diastolic Blood Pressure, Change in LDL Cholesterol | Change from Baseline at 8 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Su Youn Nam, MD, Study Director — Yuhan Corporation
Locations (1):
- Seoul National University Hospital, Seoul, South Korea

REFERENCES:
- [Derived] Oh GC, Han JK, Han KH, Hyon MS, Doh JH, Kim MH, Jeong JO, Bae JH, Kim SH, Yoo BS, Baek SH, Rhee MY, Ihm SH, Sung JH, Choi YJ, Kim SJ, Hong KS, Lee BK, Cho J, Shin ES, Rhew JY, Kim H, Kim HS. Efficacy and Safety of Fixed-dose Combination Therapy With Telmisartan and Rosuvastatin in Korean Patients With Hypertension and Dyslipidemia: TELSTA-YU (TELmisartan-rosuvaSTAtin from YUhan), a Multicenter, Randomized, 4-arm, Double-blind, Placebo-controlled, Phase III Study. Clin Ther. 2018 May;40(5):676-691.e1. doi: 10.1016/j.clinthera.2018.03.010. Epub 2018 Apr 17. PMID 29673890